CLINICAL TRIAL: NCT06153199
Title: Effectiveness and Implementation of Self-management Strategies for Low Back Pain Among Horticulture Workers
Brief Title: Self-management of Low Back Pain in Horticulture Workers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB202300756
Record Dates: First submitted 2023-11-15; First posted 2023-12-01 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Back Pain
Keywords: Self-management; Ergonomics; Horticulture workers; Video training; Guided participatory choices; Text message reminders
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-management videos (Active Comparator): Participants will review short video modules on pain self-management without medication and ergonomic work adjustment and select 1 self-management option and 1 ergonomic option to use for 10 weeks
  Interventions: Behavioral: Self-management videos
- Self-management videos + Multimodal personalized support (Experimental): Participants will review short video modules on pain self-management without medication and ergonomic work adjustment and select 1 self-management option and 1 ergonomic option to use for 10 weeks.
  Participants will use 1) checklists to guided choices for strategies based on their self-identified most difficult work activities due to pain and options that they are not using regularly, 2) review video recordings of their own work movements to assist with ergonomic problem-solving and 3) receive text message reminders
  Interventions: Behavioral: Self-management videos; Behavioral: Check lists for ergonomic options; Behavioral: Text reminders; Behavioral: Video review

INTERVENTIONS:
Behavioral: Self-management videos — Short video modules on self-management of back pain without medication and ergonomic adjustments for limiting back pain in nursery and landscape work
  Other Names: Self-management training
Behavioral: Check lists for ergonomic options — Guidance on ergonomic choices appropriate for work tasks not currently being used that are the most difficult due to back pain, using a checklist
  Arms: Self-management videos + Multimodal personalized support
Behavioral: Text reminders — Reminders to implement choices using graphics and gifs as well as motivational messages
  Other Names: Text and Graphic reminders
  Arms: Self-management videos + Multimodal personalized support
Behavioral: Video review — Participants will review videos of their movement during their most difficult work tasks to help problem solving to adjust ergonomic adjustments
  Other Names: Video feedback
  Arms: Self-management videos + Multimodal personalized support

SUMMARY:
The primary purpose of this hybrid Type II comparative effectiveness and implementation study is to compare two self-management strategies in nursery and landscape workers. This randomized pragmatic study will compare interventions with different degrees of support to determine if self-management videos plus multimodal personalized support is more effective than self-management videos alone for improving LBP among horticulture workers. Both groups will review short self-management video modules to introduce general pain concepts and the importance of managing pain without medication, risks of opioid use, self-management of pain, and simple ergonomic strategies for both groups. Both groups will choose 1 self-management strategy to manage pain at home and 1 ergonomic workplace strategy to limit pain. The video+support group will receive 1) check-list guidance, 2) review videos of their work tasks, and 3) receive text reminders to support implementation. Surveys will include instruments reflecting low back pain disability, pain, work ability, and affective or cognitive characteristics (self-efficacy, pain anxiety, depression, coping), collected at baseline, pre- and post-intervention, with follow-ups at 3- and 6-months. Workers will be videoed pre- and post-intervention for calculation of work risk and to compare any changes after the intervention. Specific aim 2 will identify contextual factors impacting engagement, adoption, effectiveness, and implementation. Interviews, focus groups, and field notes will be used to explain results and establish patterns to inform future translation.

DETAILED DESCRIPTION:
Primary dependent variables will be collected at all measurement points: pain severity, interference, and persistence, pain with specific work tasks, disability, work ability, and pain medication use. Affective or cognitive characteristics potentially impacting adoption and effectiveness (secondary dependent variables or confounders) such as coping, fear, anxiety, depression, will also be collected.The post- and follow-up survey questions will also reflect adoption, opinions of interventions, effectiveness, facilitators, and barriers.

ELIGIBILITY:
Inclusion Criteria:

Workers

1. working full time (30 hours or more per week) in physically demanding nursery or landscape work
2. currently employed or self-employed in nursery or landscape businesses
3. 18 years of age or older
4. English or Spanish speaking
5. experiencing continuous or intermittent LBP over the past 3 months

Owners, managers, supervisors

1. Owners, managers, or supervisors who meet the same inclusion criteria as workers will be eligible to participate in the training interventions as well as the supervisory roles.
2. All owners, managers, and supervisors who are willing to participate will be enrolled.

Exclusion Criteria:

Workers

1. history of major trauma, surgery, or spinal nerve blocks in the past year
2. seeking disability or workman's compensation
3. self-disclosed pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Roland Morris Disability Index | 1 year
  Disability Index for functional difficulties related to low back pain scored from 0-24 with low scores indicating lower disability
Numeric Pain Rating Severity | 1 year
  Severity of pain reported for the past week and for the 3 most difficult work activities 0=no pain, 100=worst imaginable pain, lower scores reflect lower pain
Pain Interference | 1 year
  Extent of pain interference with work activities in the past week, 0=not at all, 100=prevented working at normal level, lower scores reflect less interference
Pain persistence | 1 year
  Pain in the past 3 months reported on a 5 item scale ranging from not at all to pain every day without a break.
Pain impact | 1 year
  2 items with 5 point scale recording impact on work activities and social activities ranging from never to always, with lower scores reflecting less impact
Pain frequency | 1 year
  Number of days in the past week pain is experienced ranging from 0-7
Adoption | 1 year
  Use of the interventions reported for each work or self-management strategy selected (number of days used in the past week, how often used (never, occassionally, consistently) Higher scores and consistently are optimal
Difficulty with work tasks | 1 year
  Patient Specific Functional Scale reported for 3 most difficult work activities with subscales reported on a scale of 0= no difficulty, 100=unable to perform with the average of the 3 items used for analysis.
Work ability | 1 year
  Work Ability short form is reported on numeric rating scale from 0 (completely unable to work) to 10 able to work at your best
Use of medication and substances | 1 yeat
  Frequency of pain medication and substances for pain in past 3 months reported on a 4 item scale (never, 1-2 days, 3-4 days, 5-7 days) never is optimal. Items for alcohol, cannabis, tobacco, herbal products, acetaminophen, anti-inflammatories, muscle relaxants, opioids). Frequency of use per day on average also reported for a total estimate.

SECONDARY OUTCOMES:
Depression scale | 1 year
  Center for Epidemiology Depression Scale -Revised consists of 20 items reflecting frequency of depressive symptoms from rarely to most of the time with the total reported out of 60 with lower values as optimal
Pain anxiety Symptom Scale | 1 year
  20 item instrument with the total of items reported from never to always reported out of 50. Lower values are optimal.
Self-efficacy for Chronic Disease Management | 1 year
  PROMIS short form 8a Self-efficacy chronic disease management
Coping Skills Questionaire | 1 year
  Coping Skills Questionnaire reporting confidence to be able to work and live a normal lifestyle rated on a 6 point scale from 0=not at all confident to 5=completely confident (total reported out of 10, and 7 point scale for control over pain 0=no control, 6=completely in control. The total is reported out of 12 with higher values as optimal
Ergonomic risk | 6 months
  Rapid Ergonomic Behavioral Assessment rubric for video analysis for adjusted tasks rated out of a total of 15 indicating risk levels ranging from 1 negligible to very high

CONTACTS AND LOCATIONS:
Overall Officials: Kim Dunleavy, PT, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dunleavy K, Radunovich HL, Beneciuk JM, Hu B, Yang Y, Blythe JM, Gurka KK. Self-Management Strategies for Low Back Pain Among Horticulture Workers: Protocol for a Type II Hybrid Effectiveness-Implementation Study. JMIR Res Protoc. 2025 Jan 28;14:e64817. doi: 10.2196/64817. PMID 39874582